CLINICAL TRIAL: NCT02766582
Title: Phase II Open Label Nonrandomized Trial of the Anti PD 1 Therapy Pembrolizumab With First Line Platinum Based Chemotherapy Followed by 12 Months Pembrolizumab Monotherapy for Patients With Stage III/IV Epithelial Ovarian Cancer
Brief Title: Phase II: Pembrolizumab/Carboplatin/Taxol in Epithelial Ovary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: The Cleveland Clinic (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Denise Uyar, Associate Professor; Chief of Gynecologic Oncology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uyar 25680 IIT Merck
Record Dates: First submitted 2016-03-10; First posted 2016-05-10 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; platinum; pembrolizumab; taxane
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy combined with pembrolizumab (Experimental): Single arm study:
  Pembrolizumab IV every 21 days (200 mg) Carboplatin IV every 21 days Paclitaxel IV infusion (80 mg/m2) every 7 days for 6 cycles Followed by 12 months pembrolizumab IV every 21 days
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — IV every 21 days at 200 mg
  Other Names: Keytruda
Drug: Carboplatin — IV every 21 days
  Other Names: Paraplatin
Drug: Paclitaxel — IV infusion (80mg/m2) every 7 days for 6 cycles
  Other Names: Taxol; Onxol

SUMMARY:
Phase II single arm, open label, nonrandomized study. The aim of our study is to assess the Progression Free Survival (PFS) in suboptimally cytoreduced epithelial ovarian/ primary peritoneal/ fallopian tube cancer patients treated with the novel combination of carboplatin every 21 days (triweekly) /weekly paclitaxel IV with pembrolizumab IV followed by maintenance pembrolizumab IV.

DETAILED DESCRIPTION:
Utilization of combination standard intravenous chemotherapy with intravenous pembrolizumab (for 6 cycles) in first line treatment of patients with advanced ovarian cancer post surgery with any residual disease. This will be followed by single agent intravenous pembrolizumab (every 3 weeks) for 12 additional cycles.

ELIGIBILITY:
Inclusion Criteria:

* Have advance stage III/IV epithelial ovarian, fallopian tube or primary peritoneal cancer
* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Suboptimal cytoreductive surgery defined as any residual disease noted per operative report and/or have measurable/macroscopic disease (defined as target and/or non-target lesions) based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
* Demonstrate adequate organ function
* All screening labs should be performed within 28 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a known additional malignancy within the last 3 years, or that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study. The investigator should consult the Study Chair.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Patients with borderline ovarian tumors, recurrent epithelial ovarian/ primary peritoneal cancer/fallopian tube cancer or non-epithelial ovarian cancer are not eligible.
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10; Primary Completion 2022-05 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Uyar, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Background] Alberts DS, Green S, Hannigan EV, O'Toole R, Stock-Novack D, Anderson P, Surwit EA, Malvlya VK, Nahhas WA, Jolles CJ. Improved therapeutic index of carboplatin plus cyclophosphamide versus cisplatin plus cyclophosphamide: final report by the Southwest Oncology Group of a phase III randomized trial in stages III and IV ovarian cancer. J Clin Oncol. 1992 May;10(5):706-17. doi: 10.1200/JCO.1992.10.5.706. PMID 1569443
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964
- [Background] Swenerton K, Jeffrey J, Stuart G, Roy M, Krepart G, Carmichael J, Drouin P, Stanimir R, O'Connell G, MacLean G, et al. Cisplatin-cyclophosphamide versus carboplatin-cyclophosphamide in advanced ovarian cancer: a randomized phase III study of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 1992 May;10(5):718-26. doi: 10.1200/JCO.1992.10.5.718. PMID 1569444
- [Background] Kosary CL. FIGO stage, histology, histologic grade, age and race as prognostic factors in determining survival for cancers of the female gynecological system: an analysis of 1973-87 SEER cases of cancers of the endometrium, cervix, ovary, vulva, and vagina. Semin Surg Oncol. 1994 Jan-Feb;10(1):31-46. doi: 10.1002/ssu.2980100107. PMID 8115784
- [Background] Bristow RE, Tomacruz RS, Armstrong DK, Trimble EL, Montz FJ. Survival effect of maximal cytoreductive surgery for advanced ovarian carcinoma during the platinum era: a meta-analysis. J Clin Oncol. 2002 Mar 1;20(5):1248-59. doi: 10.1200/JCO.2002.20.5.1248. PMID 11870167
- [Background] Griffiths CT, Parker LM, Fuller AF Jr. Role of cytoreductive surgical treatment in the management of advanced ovarian cancer. Cancer Treat Rep. 1979 Feb;63(2):235-40. PMID 445502
- [Background] Hoskins WJ, McGuire WP, Brady MF, Homesley HD, Creasman WT, Berman M, Ball H, Berek JS. The effect of diameter of largest residual disease on survival after primary cytoreductive surgery in patients with suboptimal residual epithelial ovarian carcinoma. Am J Obstet Gynecol. 1994 Apr;170(4):974-9; discussion 979-80. doi: 10.1016/s0002-9378(94)70090-7. PMID 8166218
- [Background] Seidman AD, Berry D, Cirrincione C, Harris L, Muss H, Marcom PK, Gipson G, Burstein H, Lake D, Shapiro CL, Ungaro P, Norton L, Winer E, Hudis C. Randomized phase III trial of weekly compared with every-3-weeks paclitaxel for metastatic breast cancer, with trastuzumab for all HER-2 overexpressors and random assignment to trastuzumab or not in HER-2 nonoverexpressors: final results of Cancer and Leukemia Group B protocol 9840. J Clin Oncol. 2008 Apr 1;26(10):1642-9. doi: 10.1200/JCO.2007.11.6699. PMID 18375893
- [Background] Katsumata N, Yasuda M, Takahashi F, Isonishi S, Jobo T, Aoki D, Tsuda H, Sugiyama T, Kodama S, Kimura E, Ochiai K, Noda K; Japanese Gynecologic Oncology Group. Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1331-8. doi: 10.1016/S0140-6736(09)61157-0. Epub 2009 Sep 18. PMID 19767092
- [Background] Katsumata N, Yasuda M, Isonishi S, Takahashi F, Michimae H, Kimura E, Aoki D, Jobo T, Kodama S, Terauchi F, Sugiyama T, Ochiai K; Japanese Gynecologic Oncology Group. Long-term results of dose-dense paclitaxel and carboplatin versus conventional paclitaxel and carboplatin for treatment of advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer (JGOG 3016): a randomised, controlled, open-label trial. Lancet Oncol. 2013 Sep;14(10):1020-6. doi: 10.1016/S1470-2045(13)70363-2. Epub 2013 Aug 13. PMID 23948349
- [Background] Kandalaft LE, Powell DJ Jr, Singh N, Coukos G. Immunotherapy for ovarian cancer: what's next? J Clin Oncol. 2011 Mar 1;29(7):925-33. doi: 10.1200/JCO.2009.27.2369. Epub 2010 Nov 15. PMID 21079136
- [Background] Zsiros E, Tanyi J, Balint K, Kandalaft LE. Immunotherapy for ovarian cancer: recent advances and perspectives. Curr Opin Oncol. 2014 Sep;26(5):492-500. doi: 10.1097/CCO.0000000000000111. PMID 25036883
- [Background] Sato E, Olson SH, Ahn J, Bundy B, Nishikawa H, Qian F, Jungbluth AA, Frosina D, Gnjatic S, Ambrosone C, Kepner J, Odunsi T, Ritter G, Lele S, Chen YT, Ohtani H, Old LJ, Odunsi K. Intraepithelial CD8+ tumor-infiltrating lymphocytes and a high CD8+/regulatory T cell ratio are associated with favorable prognosis in ovarian cancer. Proc Natl Acad Sci U S A. 2005 Dec 20;102(51):18538-43. doi: 10.1073/pnas.0509182102. Epub 2005 Dec 12. PMID 16344461
- [Background] Zhang L, Conejo-Garcia JR, Katsaros D, Gimotty PA, Massobrio M, Regnani G, Makrigiannakis A, Gray H, Schlienger K, Liebman MN, Rubin SC, Coukos G. Intratumoral T cells, recurrence, and survival in epithelial ovarian cancer. N Engl J Med. 2003 Jan 16;348(3):203-13. doi: 10.1056/NEJMoa020177. PMID 12529460
- [Background] Hwang WT, Adams SF, Tahirovic E, Hagemann IS, Coukos G. Prognostic significance of tumor-infiltrating T cells in ovarian cancer: a meta-analysis. Gynecol Oncol. 2012 Feb;124(2):192-8. doi: 10.1016/j.ygyno.2011.09.039. Epub 2011 Oct 29. PMID 22040834
- [Background] Park A, Govindaraj C, Xiang SD, Halo J, Quinn M, Scalzo-Inguanti K, Plebanski M. Substantially modified ratios of effector to regulatory T cells during chemotherapy in ovarian cancer patients return to pre-treatment levels at completion: implications for immunotherapy. Cancers (Basel). 2012 Jun 18;4(2):581-600. doi: 10.3390/cancers4020581. PMID 24213326
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Background] Duraiswamy J, Freeman GJ, Coukos G. Therapeutic PD-1 pathway blockade augments with other modalities of immunotherapy T-cell function to prevent immune decline in ovarian cancer. Cancer Res. 2013 Dec 1;73(23):6900-12. doi: 10.1158/0008-5472.CAN-13-1550. Epub 2013 Aug 23. PMID 23975756
- [Background] Preston CC, Maurer MJ, Oberg AL, Visscher DW, Kalli KR, Hartmann LC, Goode EL, Knutson KL. The ratios of CD8+ T cells to CD4+CD25+ FOXP3+ and FOXP3- T cells correlate with poor clinical outcome in human serous ovarian cancer. PLoS One. 2013 Nov 14;8(11):e80063. doi: 10.1371/journal.pone.0080063. eCollection 2013. PMID 24244610
- [Background] Curiel TJ, Coukos G, Zou L, Alvarez X, Cheng P, Mottram P, Evdemon-Hogan M, Conejo-Garcia JR, Zhang L, Burow M, Zhu Y, Wei S, Kryczek I, Daniel B, Gordon A, Myers L, Lackner A, Disis ML, Knutson KL, Chen L, Zou W. Specific recruitment of regulatory T cells in ovarian carcinoma fosters immune privilege and predicts reduced survival. Nat Med. 2004 Sep;10(9):942-9. doi: 10.1038/nm1093. Epub 2004 Aug 22. PMID 15322536
- [Background] Hato SV, de Vries IJ, Lesterhuis WJ. STATing the importance of immune modulation by platinum chemotherapeutics. Oncoimmunology. 2012 Mar 1;1(2):234-236. doi: 10.4161/onci.1.2.18126. PMID 22720254
- [Background] Zhang L, Dermawan K, Jin M, Liu R, Zheng H, Xu L, Zhang Y, Cai Y, Chu Y, Xiong S. Differential impairment of regulatory T cells rather than effector T cells by paclitaxel-based chemotherapy. Clin Immunol. 2008 Nov;129(2):219-29. doi: 10.1016/j.clim.2008.07.013. Epub 2008 Sep 3. PMID 18771959
- [Background] Diaz Y, Tundidor Y, Lopez A, Leon K. Concomitant combination of active immunotherapy and carboplatin- or paclitaxel-based chemotherapy improves anti-tumor response. Cancer Immunol Immunother. 2013 Mar;62(3):455-69. doi: 10.1007/s00262-012-1345-y. Epub 2012 Sep 2. PMID 22941039
- [Background] Chang CL, Hsu YT, Wu CC, Lai YZ, Wang C, Yang YC, Wu TC, Hung CF. Dose-dense chemotherapy improves mechanisms of antitumor immune response. Cancer Res. 2013 Jan 1;73(1):119-27. doi: 10.1158/0008-5472.CAN-12-2225. Epub 2012 Oct 29. PMID 23108141
- [Background] Braly P, Nicodemus CF, Chu C, Collins Y, Edwards R, Gordon A, McGuire W, Schoonmaker C, Whiteside T, Smith LM, Method M. The Immune adjuvant properties of front-line carboplatin-paclitaxel: a randomized phase 2 study of alternative schedules of intravenous oregovomab chemoimmunotherapy in advanced ovarian cancer. J Immunother. 2009 Jan;32(1):54-65. doi: 10.1097/CJI.0b013e31818b3dad. PMID 19307994
- [Background] Telleria CM. Repopulation of ovarian cancer cells after chemotherapy. Cancer Growth Metastasis. 2013 Feb 18;6:15-21. doi: 10.4137/CGM.S11333. PMID 23544004
- [Background] Burger RA, Brady MF, Bookman MA, Fleming GF, Monk BJ, Huang H, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Birrer MJ, Liang SX; Gynecologic Oncology Group. Incorporation of bevacizumab in the primary treatment of ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2473-83. doi: 10.1056/NEJMoa1104390. PMID 22204724
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Seymour L, Ivy SP, Sargent D, Spriggs D, Baker L, Rubinstein L, Ratain MJ, Le Blanc M, Stewart D, Crowley J, Groshen S, Humphrey JS, West P, Berry D. The design of phase II clinical trials testing cancer therapeutics: consensus recommendations from the clinical trial design task force of the national cancer institute investigational drug steering committee. Clin Cancer Res. 2010 Mar 15;16(6):1764-9. doi: 10.1158/1078-0432.CCR-09-3287. Epub 2010 Mar 9. PMID 20215557
- [Background] Fleming TR, Rothmann MD, Lu HL. Issues in using progression-free survival when evaluating oncology products. J Clin Oncol. 2009 Jun 10;27(17):2874-80. doi: 10.1200/JCO.2008.20.4107. Epub 2009 May 4. PMID 19414672
- [Background] Basen-Engquist K, Bodurka-Bevers D, Fitzgerald MA, Webster K, Cella D, Hu S, Gershenson DM. Reliability and validity of the functional assessment of cancer therapy-ovarian. J Clin Oncol. 2001 Mar 15;19(6):1809-17. doi: 10.1200/JCO.2001.19.6.1809. PMID 11251013
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Mu CY, Huang JA, Chen Y, Chen C, Zhang XG. High expression of PD-L1 in lung cancer may contribute to poor prognosis and tumor cells immune escape through suppressing tumor infiltrating dendritic cells maturation. Med Oncol. 2011 Sep;28(3):682-8. doi: 10.1007/s12032-010-9515-2. Epub 2010 Apr 6. PMID 20373055
- [Background] Gadiot J, Hooijkaas AI, Kaiser AD, van Tinteren H, van Boven H, Blank C. Overall survival and PD-L1 expression in metastasized malignant melanoma. Cancer. 2011 May 15;117(10):2192-201. doi: 10.1002/cncr.25747. Epub 2010 Nov 29. PMID 21523733
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Garcia-Olmo DC, Dominguez C, Garcia-Arranz M, Anker P, Stroun M, Garcia-Verdugo JM, Garcia-Olmo D. Cell-free nucleic acids circulating in the plasma of colorectal cancer patients induce the oncogenic transformation of susceptible cultured cells. Cancer Res. 2010 Jan 15;70(2):560-7. doi: 10.1158/0008-5472.CAN-09-3513. Epub 2010 Jan 12. PMID 20068178
- [Background] Zhou J, Shi YH, Fan J. Circulating cell-free nucleic acids: promising biomarkers of hepatocellular carcinoma. Semin Oncol. 2012 Aug;39(4):440-8. doi: 10.1053/j.seminoncol.2012.05.013. PMID 22846861
- [Background] Kaiser J. Medicine. Keeping tabs on tumor DNA. Science. 2010 Feb 26;327(5969):1074. doi: 10.1126/science.327.5969.1074. No abstract available. PMID 20185705
- [Background] Heitzer E, Auer M, Hoffmann EM, Pichler M, Gasch C, Ulz P, Lax S, Waldispuehl-Geigl J, Mauermann O, Mohan S, Pristauz G, Lackner C, Hofler G, Eisner F, Petru E, Sill H, Samonigg H, Pantel K, Riethdorf S, Bauernhofer T, Geigl JB, Speicher MR. Establishment of tumor-specific copy number alterations from plasma DNA of patients with cancer. Int J Cancer. 2013 Jul 15;133(2):346-56. doi: 10.1002/ijc.28030. Epub 2013 Feb 13. PMID 23319339
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Murtaza M, Dawson SJ, Tsui DW, Gale D, Forshew T, Piskorz AM, Parkinson C, Chin SF, Kingsbury Z, Wong AS, Marass F, Humphray S, Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N. Non-invasive analysis of acquired resistance to cancer therapy by sequencing of plasma DNA. Nature. 2013 May 2;497(7447):108-12. doi: 10.1038/nature12065. Epub 2013 Apr 7. PMID 23563269
- [Background] Leary RJ, Sausen M, Kinde I, Papadopoulos N, Carpten JD, Craig D, O'Shaughnessy J, Kinzler KW, Parmigiani G, Vogelstein B, Diaz LA Jr, Velculescu VE. Detection of chromosomal alterations in the circulation of cancer patients with whole-genome sequencing. Sci Transl Med. 2012 Nov 28;4(162):162ra154. doi: 10.1126/scitranslmed.3004742. PMID 23197571
- [Background] Bhattacharya S, Fyfe G, Gray RJ, Sargent DJ. Role of sensitivity analyses in assessing progression-free survival in late-stage oncology trials. J Clin Oncol. 2009 Dec 10;27(35):5958-64. doi: 10.1200/JCO.2009.22.4329. Epub 2009 Oct 13. PMID 19826121
- [Background] Lakatos E. Designing complex group sequential survival trials. Stat Med. 2002 Jul 30;21(14):1969-89. doi: 10.1002/sim.1193. PMID 12111882
- [Background] Lakatos E. Sample sizes based on the log-rank statistic in complex clinical trials. Biometrics. 1988 Mar;44(1):229-41. PMID 3358991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from academic gyn oncology practice between 2016 and 2020
Groups:
- Chemotherapy Combined With Pembrolizumab: Single arm study:
  Pembrolizumab IV every 21 days (200 mg) Carboplatin IV every 21 days Paclitaxel IV infusion (80 mg/m2) every 7 days for 6 cycles Followed by 12 months pembrolizumab IV every 21 days
  Pembrolizumab: IV every 21 days at 200 mg
  Carboplatin: IV every 21 days
  Paclitaxel: IV infusion (80mg/m2) every 7 days for 6 cycles
Period: Overall Study
Arm/Group | Chemotherapy Combined With Pembrolizumab
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy Combined With Pembrolizumab
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants] — age measured in years
  Participants
    <=18 years | 0
    Between 18 and 65 years | 18
    >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] — patient age collected from electronic medical record
  years | 64 [58 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — female only
  Participants
    Female | 29
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Stage III and IV [Number; unit: units on a scale] — Stage III and IV Ovary, fallopian tube or peritoneal carcinoma with residual disease or incompletely resected disease after initial cytoreductive surgery based on imaging and surgical report. Any grade was eligible.
  units on a scale | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) of Combination Platinum Based Therapy With Anti-Programmed Death (PD)-1 Therapy Followed by Maintenance Anti-PD-1 Therapy in Patients With Epithelial Ovarian Cancer (EOC).
Description: Time to progression free survival (PFS) is the period from study entry (first dose of therapy) until disease progression, death or date of last contact.
  All patients underwent baseline computed tomographic scans prior to initiation of therapy. The residual disease information was collected from surgical operative reports as well as post operative CT scans. Treatment responses were assessed with CA 125 at each cycle of therapy. CT scans were performed post-operatively prior to initiation of systemic therapy, at the completion of combination platinum, taxane, and pembrolizumab therapy, and at the completion of maintenance pembrolizumab therapy. CT scans were also performed with increasing CA 125 or if clinically indicated per treating physician and assessments were made using response evaluation criteria in solid tumor (RECIST) criteria defined as a 20% increase in the sum of the longest diameter of target lesions, or measurable increase in non-target l
Time Frame: measured from date of completion of primary therapy to the date of the first clinical, biochemical or radiologic evidence of disease progression or death due to any cause
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Combined With Pembrolizumab
Number analyzed (Participants) | 29
months | 13.2 [11.8 to 14.7]

2. Secondary Outcome: Monitor Quality of Life During Combination Therapy and Single Agent Maintenance Therapy With Anti-PD-1 Therapy With the Functional Assessment of Cancer Therapy- Ovarian (FACT- O) Surveys at Intervals During Therapy.
Description: Each cycle is 21 days. All participants were asked to complete FACT-O surveys at baseline/ time of enrollment, at 3 months, 6 months and 18 months from initiation of therapy.
  FACT-O is a validated 26-item summary score 112 points that captures the FACT-General (FACT-G) QOL dimensions of Physical Well-Being (7 items), Functional Well-Being (7 items), and an Ovarian Cancer Subscale (12 items). FACT-0 is a survey with 39 items self administered survey. Each item is scored on 5 point Likert-type scale. The FACT-0 scoring range is from 0-44. The subscale scoring ranges for FACT-G is 0-108. The higher the total score the better the patient well-being. the outcome measure data represent FACT-G scoring as it is the section that pertains to QOL.
  https://www.facit.org/measures/FACT-O
Time Frame: Time of enrollment until 18 months from initiation of therapy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chemotherapy Combined With Pembrolizumab
Number analyzed (Participants) | 27
score on a scale
  screening | 85 [77.8 to 91]
  3 months | 88 [83 to 95]
  6 months | 83.9 [76 to 96]
  18 months | 86 [69 to 99]

3. Other Pre Specified Outcome: PD-L1 Expression in Preserved Tissue Obtained at the Time of Initial Diagnosis for Patients
Description: PD-L1 expression in preserved tissue obtained at the time of initial diagnosis for patients with suboptimally cytoreduced ovarian cancer using immunohistochemistry (IHC) of initial tumor samples and correlate with clinical outcomes of response and survival.
Time Frame: At enrollment tissue from cytoreductive surgery will be obtained from pathology blocks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 19 months
Description: AE shall mean any medical occurrence in a Study subject who is administered the Study Drug regardless of relationship with the Study Drug exists. An AE can be any unfavorable and unintended sign symptom, or disease temporally associated with the use of the Study Drug.
  SAE shall mean any untoward medical occurrence in a Study subject who is administered the Study Drug that results in death, a life-threatening drug experience, requires inpatient hospitalization or prolongation of hospitalization
Arm/Group | Chemotherapy Combined With Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 16/29
Serious Adverse Events (participants affected / at risk) | 7/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Combined With Pembrolizumab (N=29)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
encephalopathy (Nervous system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 4 (4)
acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 3 (5)
lymphopenia (Blood and lymphatic system disorders) | 4 (4)
anemia (Blood and lymphatic system disorders) | 7 (7)
nausea (Gastrointestinal disorders) | 2 (2)
heart failure (Cardiac disorders) | 1 (1)
hypothyroidism (Endocrine disorders) | 2 (2)
weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (2)
lung infection (Infections and infestations) | 1 (1)
depression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02766582/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02766582/SAP_001.pdf